CLINICAL TRIAL: NCT01282372
Title: A 2-year HRQL Observational Study Evaluating the Effect of Treatment With Adalimumab on Work Productivity and Sleep in Patients With Rheumatic Diseases in Greece
Brief Title: Greek Study on Work Productivity and Sleep in Patients With Rheumatic Diseases Treated With Adalimumab
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-179
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: Ankylosing spondylitis; Sleep; Psoriatic arthritis; Work Productivity; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with moderate to severe rheumatic disease: Participants with moderate to severe rheumatic disease (RA, PsA, or AS), who received adalimumab in accordance with approved label

SUMMARY:
Treatment with tumor necrosis factor (TNF) inhibitors, especially adalimumab, demonstrated an improvement in work productivity in participants with rheumatic diseases: rheumatoid arthritis (RA), psoriatic arthritis (PsA), and ankylosing spondylitis (AS). Limited data was available for the effect of adalimumab treatment on sleep in all three diseases (RA, PsA, and AS) and no data was available for the effect of adalimumab treatment on work productivity in PsA. This long term Health-Related Quality of Life (HRQL) observational study was conducted to evaluate the effect of treatment with adalimumab on work productivity and sleep disturbance in Greek participants with moderate to severe rheumatic diseases (RA, PsA, and AS).

DETAILED DESCRIPTION:
This was a multi-center, uncontrolled, prospective, observational study in participants with moderate to severe rheumatic disease (RA, PsA, or AS) who received adalimumab under normal clinical practice in accordance with Summary of Product Characteristics (SmPC), with or without other anti-rheumatic treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with moderate or severe active rheumatic disease, who received adalimumab under normal clinical practice in accordance with the approved local SmPC.
2. Participants who provided their consent for data collection and use by AbbVie.

Exclusion Criteria:

1. Contraindications according to the SmPC.
2. Participants who did not participate in other observational studies conducted by Abbvie.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate to severe rheumatic disease (RA, PsA, or AS), who received adalimumab in accordance with approved label, as prescribed by the physicians under normal clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theofilos Karatsourakis, MD, Study Chair — AbbVie Pharmaceuticals S.A.

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 'reason 1' and 'reason 2' for discontinuation for 'other' categories listed in participant flow is "relocation, regression of symptoms, pregnancy, and loss of insurance coverage" and "participant withdrew consent and loss of insurance coverage", respectively. AE = Adverse Event.
Period: Overall Study
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Started | 500
Completed | 421
Not Completed | 79
Not completed — Lack of Efficacy / Exacerbation | 25
Not completed — Lost to Follow-up | 23
Not completed — Withdrawal by Subject | 11
Not completed — Refer Pre-Assignment Detail for Reason 1 | 4
Not completed — Death | 1
Not completed — Presence of AE, Lack of Efficacy | 1
Not completed — Presence of AE, Regression of Symptoms | 1
Not completed — Refer Pre-Assignment Detail for Reason 2 | 1
Not completed — Adverse Event | 12

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289
  Male | 211
Employment Status [Number; unit: Participants]
  Housewife | 127
  Retired | 118
  Employee | 116
  Self-employed | 95
  Unemployed | 35
  Student | 9

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline in Work Time Missed Due to Health Problem by Disease Subgroups
Description: The 'work time missed due to health problem' was assessed using the WPAI-GHP questionnaire. WPAI-GHP is a six-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of rheumatoid diseases (RA, PsA, and AS). The 'work time missed due to health problem' was calculated based on two items: (Q2) the number of hours missed from work due to health problems in the past seven days from visit and (Q4) the number of actual work hours in the past seven days from visit. The data was calculated using the formula Q2/(Q2+Q4) and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline (Day 1) and Month 24
Population: The analysis was performed using efficacy analysis set defined as all participants in the enrolled population with an available WPAI-GHP score at the study time points.
Measure: Mean (Standard Deviation); unit: Impairment percentage
Groups:
- Participants With Moderate to Severe Rheumatic Disease - RA: Participants with moderate to severe rheumatic disease (RA), who received adalimumab in accordance with approved label
- Participants With Moderate to Severe Rheumatic Disease - PsA: Participants with moderate to severe rheumatic disease (PsA), who received adalimumab in accordance with approved label
- Participants With Moderate to Severe Rheumatic Disease - AS: Participants with moderate to severe rheumatic disease (AS), who received adalimumab in accordance with approved label
Arm/Group | Participants With Moderate to Severe Rheumatic Disease - RA | Participants With Moderate to Severe Rheumatic Disease - PsA | Participants With Moderate to Severe Rheumatic Disease - AS
Number analyzed (Participants) | 41 | 59 | 69
Impairment percentage
  Baseline | 20.7 (25.3) | 24.8 (31.1) | 17.8 (25.0)
  Change from Baseline to Month 24 (N=22, 34, 44) | -25.5 (28.6) | -21.6 (29.7) | -13.5 (26.7)

2. Primary Outcome: Mean Change From Baseline in Work Time Missed Due to Health Problem
Description: The 'work time missed due to health problem' was assessed using the Work Productivity and Activity Impairment-General Health Problem (WPAI-GHP) questionnaire. WPAI-GHP is a six-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of rheumatoid diseases (RA, PsA, and AS). The 'work time missed due to health problem' was calculated based on two items: (Q2) the number of hours missed from work due to health problems in the past seven days from visit and (Q4) the number of actual work hours in the past seven days from visit. The data was calculated using the formula Q2/(Q2+Q4) and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Impairment percentage
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 169
Impairment percentage
  Baseline | 21.0 (27.4)
  Change from Baseline to Month 24 | -18.9 (28.3)

3. Secondary Outcome: Mean Change From Baseline in Impairment While Working Due to Health Problem by Disease Subgroups
Description: The 'impairment while working due to health problem' was assessed using the WPAI-GHP questionnaire. WPAI-GHP is a six-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of rheumatoid diseases (RA, PsA, and AS). The 'impairment while working due to health problem' was calculated based on one item: (Q5) to what degree did the disease impair the productivity while working in the past seven days from visit. The item was measured on a scale from 0 (no effect) to 10 (completely prevented from doing regular activities/ working). The data was calculated using the formula Q5/10 and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Impairment percentage
Arm/Group | Participants With Moderate to Severe Rheumatic Disease - RA | Participants With Moderate to Severe Rheumatic Disease - PsA | Participants With Moderate to Severe Rheumatic Disease - AS
Number analyzed (Participants) | 40 | 57 | 69
Impairment percentage
  Baseline | 57.0 (24.4) | 49.3 (26.9) | 53.3 (26.7)
  Change from Baseline to Month 24 (N=21, 34, 43) | -50.5 (25.0) | -33.5 (30.4) | -40.0 (33.4)

4. Primary Outcome: Mean Change From Baseline in Impairment While Working Due to Health Problem
Description: as for outcome 3
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Impairment percentage
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 166
Impairment percentage
  Baseline | 52.8 (26.2)
  Change from Baseline to Month 24 | -40.0 (31.1)

5. Secondary Outcome: Mean Change From Baseline in Overall Work Impairment Due to Health Problem by Disease Subgroups
Description: The 'overall work impairment due to health problem' was assessed using the WPAI-GHP questionnaire. WPAI-GHP is a six-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of rheumatoid diseases (RA, PsA, and AS). The 'overall work impairment due to health problem' was calculated based on three items: (Q2) the number of hours missed from work due to health problems in the past seven days from visit; (Q4) the number of actual work hours in the past seven days from visit; and (Q5) to what degree did the disease impair the productivity while working past seven days from visit). The data was calculated using the formula Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)] and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Impairment percentage
Arm/Group | Participants With Moderate to Severe Rheumatic Disease - RA | Participants With Moderate to Severe Rheumatic Disease - PsA | Participants With Moderate to Severe Rheumatic Disease - AS
Number analyzed (Participants) | 40 | 53 | 66
Impairment percentage
  Baseline | 62.3 (25.1) | 53.9 (27.4) | 58.3 (27.6)
  Change from Baseline to Month 24 (N=21, 31, 42) | -55.2 (26.0) | -40.6 (32.7) | -47.1 (32.1)

6. Primary Outcome: Mean Change From Baseline in Overall Work Impairment Due to Health Problem
Description: as for outcome 5
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Impairment percentage
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 159
Impairment percentage
  Baseline | 57.8 (26.9)
  Change from Baseline to Month 24 | -46.8 (31.2)

7. Secondary Outcome: Mean Change From Baseline in Overall Activity Impairment Due to Health Problem by Disease Subgroups
Description: The 'overall activity impairment due to health problem' was assessed using the WPAI-GHP questionnaire. WPAI-GHP is a six-item participant-assessed questionnaire used to assess work and activity impairment due to symptoms of rheumatoid diseases (RA, PsA, and AS). The 'overall activity impairment due to health problem' was calculated based on one item: (Q6) to what degree did the disease impair the ability to do regular activities in the past seven days from visit. The item was measured on a scale from 0 (no effect) to 10 (completely prevented from doing regular activities/working). The data was calculated using the formula Q6/10 and converted to percent. Data are presented as impairment percentage, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Impairment percentage
Arm/Group | Participants With Moderate to Severe Rheumatic Disease - RA | Participants With Moderate to Severe Rheumatic Disease - PsA | Participants With Moderate to Severe Rheumatic Disease - AS
Number analyzed (Participants) | 184 | 166 | 150
Impairment percentage
  Baseline | 64.5 (24.4) | 59.4 (23.3) | 62.1 (24.9)
  Change from Baseline to Month 24 (N=155, 139, 127) | -47.5 (28.2) | -45.8 (26.1) | -47.6 (28.5)

8. Primary Outcome: Mean Change From Baseline in Overall Activity Impairment Due to Health Problem
Description: as for outcome 7
Time Frame: Baseline (Day 1) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Impairment percentage
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 500
Impairment percentage
  Baseline | 62.1 (24.2)
  Change from Baseline to Month 24 | -47.0 (27.6)

9. Secondary Outcome: Mean Disease Activity Score 28 (DAS28)
Description: The DAS28, a combined index that measured rheumatoid arthritis disease activity, was calculated based on: (1) the number of tender joints among 28 joints evaluated; (2) the number of swollen joints among 28 joints evaluated; (3) general health evaluated by a visual analog scale (VAS); (4) erythrocyte sedimentation rate (ESR); and (5) C-reactive protein (CRP). The DAS28 scores ranged from 0 (no disease activity) to 10 (maximal disease activity); decrease in DAS28 scores indicate improvement of disease. The DAS28 score less than or equal to 2.6 is defined as clinical remission. Data are presented as mean DAS28 score +/- standard deviation.
Time Frame: Baseline (Day 1), Month 3, Month 6, Month 12, Month 18, and Month 24
Population: The analysis was performed using efficacy analysis set defined as all participants in the enrolled population with an available DAS28 score at the study time points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Participants With Moderate to Severe Rheumatic Disease: Participants with moderate to severe rheumatic disease (RA), who received adalimumab in accordance with approved label
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 184
Scores on a scale
  Baseline | 5.95 (1.16)
  Month 3 (N= 179) | 4.05 (1.35)
  Month 6 (N=175) | 3.39 (1.26)
  Month 12 (N=164) | 3.08 (1.27)
  Month 18 (N=160) | 2.90 (1.21)
  Month 24 (N=153) | 2.72 (1.28)

10. Secondary Outcome: Mean Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The HAQ-DI was a participant-reported questionnaire that measured quality of life in terms of physical function of participants with rheumatoid arthritis. It consisted of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past seven days using the following response categories (score): without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). The scores on each task were summed and averaged to provide an overall score from 0 to 3, where 0-1 represented mild disability and 2-3 represented severe disability. Data are presented as mean HAQ-DI score +/- standard deviation.
Time Frame: Baseline (Day 1), Month 3, Month 6, Month 12, Month 18, and Month 24
Population: The analysis was performed using efficacy analysis set defined as all participants in the enrolled population with an available HAQ-DI score at the study time points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 181
Scores on a scale
  Baseline | 1.60 (0.61)
  Month 3 (N=179) | 0.98 (0.62)
  Month 6 (N=176) | 0.77 (0.55)
  Month 12 (N=164) | 0.65 (0.54)
  Month 18 (N=159) | 0.58 (0.55)
  Month 24 (N=153) | 0.51 (0.53)

11. Secondary Outcome: Mean Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score
Description: The BASDAI was a six question, participant-reported measure of overall disease activity that probed the level of fatigue, neck/back/hip pain, peripheral joint swelling and pain, localized tenderness, as well as morning stiffness severity and duration. The mean measurement (score) of questions 5 and 6 is added to the scores from questions 1 to 4 and divided by 5 to calculate the total BASDAI score. It was scored on a numerical rating scale that ranged from 0 (no symptoms) to 10 (severe symptoms), higher scores indicating severe disability due to AS disease. Data are presented as mean total BASDAI score +/- standard deviation.
Time Frame: Baseline (Day 1), Month 3, Month 6, Month 12, Month 18, and Month 24
Population: The analysis was performed using efficacy analysis set defined as all participants in the enrolled population with an available BASDAI score at the study time points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Participants With Moderate to Severe Rheumatic Disease: Participants with moderate to severe rheumatic disease (AS), who received adalimumab in accordance with approved label
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 146
Scores on a scale
  Baseline | 5.75 (1.67)
  Month 3 | 3.34 (1.71)
  Month 6 (N=138) | 2.51 (1.55)
  Month 12 (N=130) | 2.05 (1.48)
  Month 18 (N=125) | 1.69 (1.24)
  Month 24 (N=125) | 1.50 (1.28)

12. Secondary Outcome: Mean Psoriatic Arthritis Response Criteria (PsARC) Score
Description: As the patient and physician global assessments were performed using a 0-100 VAS scale instead of the 5 point Likert scale, the PsARC score could not be calculated, although data on joint pain and swelling were collected. Hence, the psoriatic arthritis disease activity was evaluated by the percentage of patients with tender and swollen joints, acute phase reactants (ESR and CRP), and VAS Score (patient and physician). Data are reported under outcome measures 13 through 16.
Time Frame: Baseline (Day 1), Month 3, Month 6, Month 12, Month 18, and Month 24
Population: The PsARC score was not assessed in this study.
Arm/Group | Participants With Moderate to Severe Rheumatic Disease - PsA
Number analyzed (Participants) | 0

13. Secondary Outcome: Percentage of Participants With Tender Joint Count (TJC) and Swollen Joint Count (SJC) Greater Than Zero
Description: Joints (68 or 66) were assessed by pressure and joint manipulation on physical examination for TJC or SJC, respectively. Both joint tenderness and swelling were classified as present ("1"), absent ("0"), replaced ("9"), or no assessment ("NA"). The total TJC or SJC was derived as the sum of the tender and swollen joints; the range for TJC and SJC were 0 - 68 and 0 - 66, respectively with higher scores indicated worse conditions. Data are presented as percentage of participants with TJC and SJC.
Time Frame: Baseline (Day 1), Month 3, Month 6, Month 12, Month 18, and Month 24
Population: The analysis was performed using efficacy analysis set defined as all participants in the enrolled population with evaluable data at the study time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Moderate to Severe Rheumatic Disease - PsA
Number analyzed (Participants) | 166
Percentage of participants
  TJC at Baseline | 98.8
  TJC at Month 3 (N=163) | 72.4
  TJC at Month 6 (N=155) | 48.4
  TJC at Month 12 (N=147) | 34.0
  TJC at Month 18 (N=144) | 32.6
  TJC at Month 24 (N=139) | 28.1
  SJC at Baseline | 91.0
  SJC at Month 3 (N=163) | 52.8
  SJC at Month 6 (N=155) | 32.3
  SJC at Month 12 (N=147) | 26.5
  SJC at Month 18 (N=144) | 28.5
  SJC at Month 24 (N=139) | 17.3

14. Secondary Outcome: Mean Erythrocyte Sedimentation Rate (ESR)
Description: Plasma concentrations were assessed to evaluate ESR, a marker of systemic inflammation that provided insights into the overall anti-inflammatory effect of rheumatologic therapies. Data are presented as mean ESR value in millimeters per hour (mm/hr) ± standard deviation.
Time Frame: Baseline (Day 1), Month 3, Month 6, Month 12, Month 18, and Month 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Participants With Moderate to Severe Rheumatic Disease - PsA
Number analyzed (Participants) | 158
mm/hr
  Baseline | 40.2 (22.1)
  Month 3 (N=157) | 25.3 (15.4)
  Month 6 (N=150) | 21.7 (16.3)
  Month 12 (N=146) | 18.5 (13.3)
  Month 18 (N=140) | 17.6 (12.6)
  Month 24 (N=137) | 16.2 (11.5)

15. Secondary Outcome: Mean Plasma Concentrations of C-Reactive Protein (CRP)
Description: Plasma concentrations were assessed to evaluate CRP, a marker of systemic inflammation that provided insights into the overall anti-inflammatory effect of rheumatologic therapies. Data are presented as mean CRP value in milligrams per liter (mg/L) ± standard deviation.
Time Frame: Baseline (Day 1), Month 3, Month 6, Month 12, Month 18, and Month 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Participants With Moderate to Severe Rheumatic Disease - PsA
Number analyzed (Participants) | 150
mg/L
  Baseline | 9.94 (13.93)
  Month 3 (N=144) | 5.05 (9.48)
  Month 6 (N=140) | 3.26 (6.49)
  Month 12 (N=141) | 1.94 (3.05)
  Month 18 (N=137) | 1.99 (3.60)
  Month 24 (N=133) | 1.91 (4.16)

16. Secondary Outcome: Mean Visual Analogue Scale (VAS) Score
Description: The VAS score assessed by participants (pt) and physicians (ph) was used to determine the pain due to psoriatic arthritis in the past week. The level of pain was measured in millimeters (mm) on a 100 mm horizontal line. The score ranged from 0 (no pain) to 100 (severe pain). Data are presented as mean VAS score +/- standard deviation.
Time Frame: Baseline (Day 1), Month 3, Month 6, Month 12, Month 18, and Month 24
Population: The analysis was performed using efficacy analysis set defined as all participants in the enrolled population with an available VAS score at the study time points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Participants With Moderate to Severe Rheumatic Disease: Participants with moderate to severe rheumatic disease (PsA), who received adalimumab in accordance with approved label
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 166
Scores on a scale
  VAS pt at Baseline | 65.80 (16.90)
  VAS pt at Month 3 (N=163) | 32.00 (19.40)
  VAS pt at Month 6 (N=155) | 21.90 (18.20)
  VAS pt at Month 12 (N=147) | 15.10 (13.90)
  VAS pt at Month 18 (N=144) | 14.10 (13.20)
  VAS pt at Month 24 (N=139) | 12.00 (13.60)
  VAS ph at Baseline | 62.55 (16.70)
  VAS ph at Month 3 (N=163) | 29.30 (19.40)
  VAS ph at Month 6 (N=155) | 19.67 (17.40)
  VAS ph at Month 12 (N=147) | 14.20 (15.10)
  VAS ph at Month 18 (N=144) | 12.75 (12.10)
  VAS ph at Month 24 (N=139) | 11.31 (13.90)

17. Secondary Outcome: Mean Sleep Disturbance Subscale Score
Description: The Medical Outcome Study (MOS) sleep scale was a 12-item, participant-reported, non-disease-specific measure related to sleep that yielded 7 subscales (4-item sleep disturbance, 2-item sleep adequacy, 1-item quantity of sleep, 3-item somnolence, 1-item snoring, 1-item shortness of breath, and 9-item overall sleep problems index). Only sleep disturbance subscale was assessed by calculating the average of the 4-items with total score ranging from 0 to 100 (higher scores indicating greater sleep disturbance). Data are presented as mean score on a scale +/- standard deviation.
Time Frame: Baseline (Day 1), Month 3, Month 6, Month 12, Month 18, and Month 24
Population: The analysis was performed using safety analysis set defined as all participants who received at least one dose of adalimumab.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Number analyzed (Participants) | 500
Scores on a scale
  Baseline | 50.9 (23.6)
  Month 3 (N=492) | 30.3 (18.0)
  Month 6 (N=472) | 23.4 (16.7)
  Month 12 (N=446) | 19.7 (16.9)
  Month 18 (N=432) | 18.3 (15.7)
  Month 24 (N=421) | 16.6 (15.6)

ADVERSE EVENTS:
Time Frame: Up to 2 years from signing of informed consent
Description: The occurrence, type, severity, and relationship of adverse events to adalimumab were assessed.
Arm/Group | Participants With Moderate to Severe Rheumatic Disease
Serious Adverse Events (participants affected / at risk) | 33/500
Other Adverse Events (participants affected / at risk) | 158/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Moderate to Severe Rheumatic Disease (N=500)
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Anaphylactic shock (Immune system disorders) | 1
Rash pustular (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
VIIth nerve injury (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Choroid plexus papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypoaesthesia (Nervous system disorders) | 1
Hypoglycaemic coma (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Moderate to Severe Rheumatic Disease (N=500)
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Sturge-Weber syndrome (Congenital, familial and genetic disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Drug effect incomplete (General disorders) | 1
Drug ineffective (General disorders) | 24
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 3
Peripheral swelling (General disorders) | 1
Polyp (General disorders) | 1
Pyrexia (General disorders) | 10
Hypertransaminasemia (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 3
Bronchopneumonia (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Metabolism and nutrition disorders (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 13
Respiratory tract infection viral (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 6
Vaginal infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Drug dose omission (Injury, poisoning and procedural complications) | 1
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Blood glucose increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Drug specific antibody present (Investigations) | 1
Glycosylated hemoglobin increased (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 11
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Burning sensation (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Normal newborn (Pregnancy, puerperium and perinatal conditions) | 1
Anxiety disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 1
Albuminuria (Renal and urinary disorders) | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 3
Purpura (Skin and subcutaneous tissue disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.